CLINICAL TRIAL: NCT06030947
Title: Tunnel Surgery Combined With a Micro Connective Tissue Graft for the Treatment of Multiple Adjacent Gingival Recession Defects: a Multi-center Randomized Controlled Clinical Trial.
Brief Title: Effectiveness of Micro Connective Tissue Graft for Treatment of Multiple Adjacent Gingival Recession Defects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OCarcuac-microCTG
Record Dates: First submitted 2023-09-03; First posted 2023-09-11 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Gingival Recession, Localized
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connective Tissue Graft (Active Comparator): A mucogingival surgery where a conventional connective tissue graft harvested from the palate is placed on a recipient site prepared for modified coronally advanced tunnel and sutured to cover multiple adjacent gingival recession defects.
  Interventions: Procedure: Coronally Advanced Flap combined with a Connective Tissue Graft
- Micro Connective Tissue Graft (Experimental): A mucogingival surgery where multiple micro connective tissue graft harvested from the palate are placed on a recipient site prepared for modified coronally advanced tunnel and sutured to cover multiple adjacent gingival recession defects.
  Interventions: Procedure: Coronally Advanced Flap combined with micro Connective Tissue Graft; Device: Division of the Connective Tissue Graft into multiple micro Connective Tissue Grafts

INTERVENTIONS:
Procedure: Coronally Advanced Flap combined with a Connective Tissue Graft — Multiple adjacent gingival recession defects will be covered by coronally advanced flap combined with a connective tissue graft harvested from the palate.
  Arms: Connective Tissue Graft
Procedure: Coronally Advanced Flap combined with micro Connective Tissue Graft — Multiple adjacent gingival recession defects will be covered by coronally advanced flap combined with multiple micro connective tissue graft harvested from the palate.
  Arms: Micro Connective Tissue Graft
Device: Division of the Connective Tissue Graft into multiple micro Connective Tissue Grafts — The harvested connective tissue graft is divided in multiple micro connective tissue grafts with a scalpel blade before being placed on the recipient site.
  Arms: Micro Connective Tissue Graft

SUMMARY:
The objective of this project is to evaluate 1-year outcomes of treatment of MAGRD using a modified coronally advanced tunnel technique (MCAT) with either conventional CTG (control group) or micro-CTG (test group).

DETAILED DESCRIPTION:
Gingival recession defects (GRD) present as a partial exposure of the root surface resulting from gingival margin displacement apical to the cemento-enamel junction (CEJ). A variety of surgical methods have been reported to reestablish root coverage, including tunneling techniques and coronally and laterally advanced flaps. As the presence of thin gingival tissues is one of the predisposing factors for GRD, the adjuvant use of subepithelial connective tissue grafts (CTGs) during the surgical correction is often considered. CTGs are thought to contribute to phenotype modification and stability of treatment outcomes and studies have indicated favorable esthetic results and high degrees of root coverage (documented range: 69% to 97%). The procedure does, however, require a suitable donor site. When multiple adjacent teeth exhibit GRDs, the preferred surgical approach should offer the greatest possible root coverage, while limiting drawbacks (i.e., patient morbidity, esthetic problems). Thus, one of the challenges related to coverage of multiple GRDs is the scarcity of donor tissue. In cases when large CTGs are required, additional surgical procedures may even be necessary. As an alternative, a modification of the harvested CTG into multiple "micro-CTGs" is proposed for the treatment of multiple adjacent GRDs (MAGRD). In the present study, the effectiveness and predictability of micro-CTGs will be evaluated in direct comparison to conventional CTGs.

The investigators hypothesise that no statistically significant differences will be observed in terms of % root coverage (primary outcome) and patient satisfaction at 12 months (non-inferiority).

The investigators hypothesise that subjects in the test group (micro-CTG) will report significantly lower morbidity at 1 and 2 weeks post-surgery when compared to controls (superiority).

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years,
* systemically healthy,
* presenting with a minimum of 4 and a maximum of 6 adjacent RT1/RT2 recessions, located in the maxilla or mandible with an apico-coronal extension (i.e. recession depth) of ≥2 mm,
* Full-Mouth Plaque Score (FMPS) <20%,
* Full-Mouth Bleeding Score (FMBS) <20%.

Exclusion Criteria:

* pregnancy or lactation,
* tobacco smoking,
* uncontrolled medical condition,
* medication that can affect gingival conditions.
* thick phenotype,
* severe tooth malpositioning,
* uncorrected trauma from toothbrushing,
* a previous history of root coverage procedures
* the presence of furcation defects.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Mean mid-facial recession coverage (mRC) | up to 1 year
  Percentage of the exposed tooth root covered after surgical intervention

SECONDARY OUTCOMES:
Complete Root Coverage (CRC) | up to 1 year
  Frequency of complete root coverage
Changes of Keratinized Tissue Width (KTW) | up to 1 year
  Measured as the distance from the muco-gingival-junction to the gingival margin
Changes of Gingival Thickness (GT) | up to 1 year
  Measured 3 mm apically from the free gingival margin at the mid-buccal aspect of the tooth
Patient Morbidity | up to 2 weeks
  Measured with Visual Analogue Scale (VAS), which consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be')
Patient Satisfaction | up to 1 year
  Measured with Visual Analogue Scale (VAS), which consists of a 10cm line, with two end points representing 0 ('not satisfied') and 10 ('satisfied as much as it could possibly be')

CONTACTS AND LOCATIONS:
Overall Officials: Jan Derks, DDS, PhD, Study Chair — Goteborg University
Locations (1):
- Confident Dubai Palm, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Consensus report. Mucogingival therapy. Ann Periodontol. 1996 Nov;1(1):702-6. doi: 10.1902/annals.1996.1.1.702. No abstract available. PMID 9118277
- [Result] Cairo F. Periodontal plastic surgery of gingival recessions at single and multiple teeth. Periodontol 2000. 2017 Oct;75(1):296-316. doi: 10.1111/prd.12186. PMID 28758301
- [Result] Tonetti MS, Jepsen S; Working Group 2 of the European Workshop on Periodontology. Clinical efficacy of periodontal plastic surgery procedures: consensus report of Group 2 of the 10th European Workshop on Periodontology. J Clin Periodontol. 2014 Apr;41 Suppl 15:S36-43. doi: 10.1111/jcpe.12219. PMID 24640999
- [Result] Cairo F, Nieri M, Pagliaro U. Efficacy of periodontal plastic surgery procedures in the treatment of localized facial gingival recessions. A systematic review. J Clin Periodontol. 2014 Apr;41 Suppl 15:S44-62. doi: 10.1111/jcpe.12182. PMID 24641000
- [Result] Graziani F, Gennai S, Roldan S, Discepoli N, Buti J, Madianos P, Herrera D. Efficacy of periodontal plastic procedures in the treatment of multiple gingival recessions. J Clin Periodontol. 2014 Apr;41 Suppl 15:S63-76. doi: 10.1111/jcpe.12172. PMID 24641002
- [Result] Ronco V, Dard M. A novel suturing approach for tissue displacement within minimally invasive periodontal plastic surgery. Clin Case Rep. 2016 Jul 23;4(8):831-7. doi: 10.1002/ccr3.582. eCollection 2016 Aug. PMID 27525096